CLINICAL TRIAL: NCT00381186
Title: Impact of 3-year Lifestyle Intervention on Postprandial Glucose Metabolism: the SLIM Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NWO 2200.0139; ZonMW 940-35-034; DFN 98.901 and 2000.00.020
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2006-09

CONDITIONS: Impaired Glucose Tolerance; Type 2 Diabetes
Keywords: impaired glucose tolerance; type 2 diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Diet

INTERVENTIONS:
Behavioral: diet- and exercise intervention

SUMMARY:
To evaluate the effect of a 3-year diet- and exercise lifestyle intervention, based on general public health recommendations, on glucose tolerance, insulin resistance and metabolic cardiovascular risk factors in Dutch subjects with impaired glucose tolerance (IGT).

DETAILED DESCRIPTION:
Objective To evaluate the effect of a 3-year diet- and exercise lifestyle intervention, based on general public health recommendations, on glucose tolerance, insulin resistance and metabolic cardiovascular risk factors in Dutch subjects with impaired glucose tolerance (IGT).

Research design and methods 147 IGT subjects (75 male, 72 female) were randomized to the intervention group (INT) or control group (CON). 106 subjects (52 INT, 54 CON) completed 3 years of intervention. Annually, glucose, insulin and FFA concentrations were determined during fasting and after an oral glucose tolerance test, in addition to measurements of body weight, serum lipids, blood pressure and maximal aerobic capacity.

ELIGIBILITY:
Inclusion Criteria:

* caucasion,age 40-70, mean 2hr glucose 7.8-12.5 mmol/l, mean fasting blood glucose below 7.8

Exclusion Criteria:

* known type 2 diabetes, mean 2hr glucose >12.5 mmol/l, mean fasting blood glucose > 7.8 mmol/l, chronic illness that makes 5-year survival improbable, interferes with glucose tolerance or makes participation in a lifestyle intervention impossible, medication known to interfere with glucose tolerance, participation in a vigorous exercise and/or diet program

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1999-02; Study Completion 2006-06

PRIMARY OUTCOMES:
2-hour glucose levels
insulin resistance

SECONDARY OUTCOMES:
adherence
type 2 diabetes
dietary intake change
exercise change

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, PhD, Principal Investigator — Maastricht University, Department of Human Biology; Wim HM Saris, PhD, Study Chair — Maastricht University, Department of Human Biology

REFERENCES:
- [Derived] den Boer AT, Herraets IJ, Stegen J, Roumen C, Corpeleijn E, Schaper NC, Feskens E, Blaak EE. Prevention of the metabolic syndrome in IGT subjects in a lifestyle intervention: results from the SLIM study. Nutr Metab Cardiovasc Dis. 2013 Nov;23(11):1147-53. doi: 10.1016/j.numecd.2012.12.005. Epub 2013 Feb 23. PMID 23462149
- [Derived] Penn L, White M, Lindstrom J, den Boer AT, Blaak E, Eriksson JG, Feskens E, Ilanne-Parikka P, Keinanen-Kiukaanniemi SM, Walker M, Mathers JC, Uusitupa M, Tuomilehto J. Importance of weight loss maintenance and risk prediction in the prevention of type 2 diabetes: analysis of European Diabetes Prevention Study RCT. PLoS One. 2013;8(2):e57143. doi: 10.1371/journal.pone.0057143. Epub 2013 Feb 25. PMID 23451166
- [Derived] Roumen C, Feskens EJ, Corpeleijn E, Mensink M, Saris WH, Blaak EE. Predictors of lifestyle intervention outcome and dropout: the SLIM study. Eur J Clin Nutr. 2011 Oct;65(10):1141-7. doi: 10.1038/ejcn.2011.74. Epub 2011 May 18. PMID 21587283